CLINICAL TRIAL: NCT04108663
Title: Lasting Amelioration of Deficient Cognitive Control by Transcranial Direct Current Stimulation (tDCS)-Enhanced Training
Brief Title: Supporting Cognitive Control Training With tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Christian Plewnia, MD, Doctor of Psychiatry and Psychotherapy, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GCBS-WP4
Record Dates: First submitted 2019-09-17; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Cognitive Control
Keywords: Brain stimulation; Cognitive training; Cognition; Cognitive enhancement; Transcranial direct current stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (9):
- Sham (Sham Comparator): Sham tDCS (ramp up and ramp down of electrical current before as well as after task performance to elicit physical sensations similar to verum tDCS)
  Interventions: Behavioral: Effect of tDCS on cognitive control task performance
- L1A (Active Comparator): Active tDCS
  * laterality: left PFC (F3; second electrode placed on deltoid muscle of the opposing arm)
  * intensity: of 1 mA
  * polarity: anodal
  Interventions: Behavioral: Effect of tDCS on cognitive control task performance
- R1A (Active Comparator): Active tDCS
  * laterality: right PFC (F4; second electrode placed on deltoid muscle of the opposing arm)
  * intensity: of 1 mA
  * polarity: anodal
  Interventions: Behavioral: Effect of tDCS on cognitive control task performance
- L2A (Active Comparator): Active tDCS
  * laterality: left PFC (F3; second electrode placed on deltoid muscle of the opposing arm)
  * intensity: of 2 mA
  * polarity: anodal
  Interventions: Behavioral: Effect of tDCS on cognitive control task performance
- R2A (Active Comparator): Active tDCS
  * laterality: right PFC (F4; second electrode placed on deltoid muscle of the opposing arm)
  * intensity: of 2 mA
  * polarity: anodal
  Interventions: Behavioral: Effect of tDCS on cognitive control task performance
- L1C (Active Comparator): Active tDCS
  * laterality: left PFC (F3; second electrode placed on deltoid muscle of the opposing arm)
  * intensity: of 1 mA
  * polarity: cathodal
  Interventions: Behavioral: Effect of tDCS on cognitive control task performance
- R1C (Active Comparator): Active tDCS
  * laterality: right PFC (F4; second electrode placed on deltoid muscle of the opposing arm)
  * intensity: of 1 mA
  * polarity: cathodal
  Interventions: Behavioral: Effect of tDCS on cognitive control task performance
- L2C (Active Comparator): Active tDCS
  * laterality: left PFC (F3; second electrode placed on deltoid muscle of the opposing arm)
  * intensity: of 2 mA
  * polarity: cathodal
  Interventions: Behavioral: Effect of tDCS on cognitive control task performance
- R2C (Active Comparator): Active tDCS
  * laterality: right PFC (F4; second electrode placed on deltoid muscle of the opposing arm)
  * intensity: of 2 mA
  * polarity: cathodal
  Interventions: Behavioral: Effect of tDCS on cognitive control task performance

INTERVENTIONS:
Behavioral: Effect of tDCS on cognitive control task performance — Added verum or sham tDCS while working on a cognitive control task.

SUMMARY:
Cognitive control (CC) is an important prerequisite for goal-directed behaviour and often associated with dysfunctional prefrontal activity within the cortex. This can be ameliorated by non-invasive brain stimulation. In this randomised single-blind study we compare effects of transcranial direct current stimulation (tDCS) on CC in healthy subjects. The study includes 162 subjects who undergo a two-week (six sessions) training of cognitive control (adaptive paced auditory serial addition task, PASAT) supported by tDCS. Subjects are randomised to receive either concurrent anodal, cathodal, or sham tDCS with an intensity of 1 mA or 2 mA of their left (F3) or right (F4) PFC, resulting in eight stimulation groups. Stimulation effects on performance changes are compared to a sham control group.Changes in Affective state are measured by the positive and negative affect schedule (PANAS), possible transfer effects are assessed by the Eriksen Flanker task. Stability of effects is measured up to three months after the last intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Right-handed (assessed by Edinburgh Handedness Inventory)
* No other concurrent brain stimulation during participation
* Proficient in German (min. CEFR level B)
* Ability to strictly adhere to study timeline

Exclusion Criteria:

* Diagnosed neurological illnesses
* Diagnosed psychiatric disorders
* Achromatopsia
* Metallic implants / tattoos on or near electrode sites
* Consumption of tobacco to an equivalent of ten or more cigarettes per day
* Prior participation in experiments involving the PASAT

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 2 to 14 weeks
  Changes in performance in the PASAT (as assessed by number of correct trials within each PASAT session) due to the various tDCS interventions. All eight interventions will be compared to the sham group. Cognitive performance is modified by tDCS, which is applied through a multi-channel stimulator (DC-Stimulator MC, NeuroConn GmbH, Ilmenau, Germany; software version 1.3.8; two rectangular rubber electrodes (5 x 7 cm)).

SECONDARY OUTCOMES:
Affective state | 2 weeks
  Changes in affective state over the course of the experiment (assessed by the positive and negative affect schedule (PANAS) questionnaire). Scores are calculated for negative and positive affect separately, by summing up the respective answers.
Transfer effect | 3 weeks
  Transfer effects in the Eriksen Flanker task (assessed through mean reaction times). Means are calculated for congruent, incongruent, and neutral trials respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Plewnia, MD, Principal Investigator — University of Tübingen, Department of Psychiatry and Psychotherapy
Locations (1):
- University of Tübingen, Department of Psychiatry and Psychotherapy, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weller S, Derntl B, Plewnia C. Sex matters for the enhancement of cognitive training with transcranial direct current stimulation (tDCS). Biol Sex Differ. 2023 Nov 2;14(1):78. doi: 10.1186/s13293-023-00561-4. PMID 37919761
- [Derived] Weller S, Nitsche MA, Plewnia C. Enhancing cognitive control training with transcranial direct current stimulation: a systematic parameter study. Brain Stimul. 2020 Sep-Oct;13(5):1358-1369. doi: 10.1016/j.brs.2020.07.006. Epub 2020 Jul 18. PMID 32687899